CLINICAL TRIAL: NCT06379906
Title: The Association Between Upper Extremity Muscle Strength, Balance and Functional Skills in Children With Duchenne Muscular Dystrophy
Brief Title: Upper Extremity Muscle Strength, Balance and Functional Skills in DMD
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Collaborators: Biruni University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Gülsena Utku, Research Assistant, Halic University
Other Study IDs: DMD, UE and Balance
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: duchenne muscular dystrophy; upper extremity; balance; functional skills
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Baseline assessment

SUMMARY:
This study aims to examine the relationship between upper extremity muscle strength, balance and functional skills of children with DMD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with DMD by a child neurologist and confirmed by genetic test results,
* were at Level 1-4 according to Brooke Lower Extremity Functional Classification (able to ambulate independently and get up from a chair)
* had cooperation with the researchers

Exclusion Criteria:

* had undergone a surgical operation in the last 6 months
* had contractures that would affect functional activities

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants who applied to the Child Neurology outpatient clinic of Istanbul University, Istanbul Faculty of Medicine, Department of Child Health and Diseases
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Muscle Strength Measurements | one time (baseline)
Trunk Control Measurement Scale | one time (baseline)
Functional Reach Test | one time (baseline)
Timed Up & Go Test | one time (baseline)

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory | one time (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: GÜLSENA UTKU UMUT, Principal Investigator — HALİÇ UNİVERSİTY
Locations (1):
- Haliç University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided